CLINICAL TRIAL: NCT03751098
Title: A Multi-Center, Double-Masked, Placebo-Controlled, Phase 3 Study of the Safety and Efficacy of Fixed Combination Phenylephrine 2.5%-Tropicamide 1% Ophthalmic Solution Administered With a Microdose Dispenser for Dilation of the Pupil
Brief Title: Safety and Efficacy of Phenylephrine 2.5%-Tropicamide 1% Microdose Ophthalmic Solution for Pupil Dilation
Acronym: MIST-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: EYN-MYD-TP-32
Record Dates: First submitted 2018-11-14; First posted 2018-11-23 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-01

CONDITIONS: Mydriasis
MeSH Terms: conditions — Mydriasis | interventions — Tropicamide

STUDY DESIGN:
Intervention Model Description: This trial was a double-masked, placebo-controlled, cross-over superiority study evaluating the efficacy of the fixed combination drug vs. placebo. All participants in the trial were to receive each treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: There were no differences in the presentation of study treatment administered and all study personnel conducting ophthalmic assessments after study treatment administration were masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1-TR/PE, 2-Placebo, 3-Placebo (Other): Participants were dosed once at 3 separate clinic visits in accordance with this sequence. Each participant received 2 sprays of the designated treatment in each eye.
  Interventions: Drug: Tropicamide/Phenylephrine ophthalmic solution (TR/PE); Drug: Placebo
- 1-Placebo, 2-Placebo, 3-TR/PE (Other): Participants were dosed once at 3 separate clinic visits in accordance with this sequence. Each participant received 2 sprays of the designated treatment in each eye.
  Interventions: Drug: Tropicamide/Phenylephrine ophthalmic solution (TR/PE); Drug: Placebo

INTERVENTIONS:
Drug: Tropicamide/Phenylephrine ophthalmic solution (TR/PE) — Tropicamide 1%/phenylephrine 2.5% ophthalmic solution administered with the Optejet microdose dispenser
  Other Names: Mydcombi
Drug: Placebo — Eyewash administered with the Optejet microdose dispenser

SUMMARY:
This study evaluated pupil dilation after administration of fixed combination tropicamide-phenylephrine (TR/PH) vs. placebo. Participants attended 3 visits. At each visit, after baseline measurements, either the study drug or placebo was administered to both eyes, then pupil dilation and safety assessments were performed at specific time intervals.

DETAILED DESCRIPTION:
Volunteer participants were screened for study eligibility during a Screening Visit and enrolled after signing the study-specific informed consent form. Subjects meeting all inclusion/exclusion criteria were scheduled for 3 treatment visits, which were at least 2 days, but no more than 7 days apart. At each treatment visit, baseline measurements were taken, then either the study drug or placebo was administered to both eyes. Afterwards, efficacy and safety assessments were performed at 20, 35, 50, 65, 80, 120, and 180 minutes. Participants' treatment assignments for each treatment visit were equally randomized using 1 of 2 sequences - ABB or BAA, where A was the study drug and B was the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written consent and return for all study visits
* Photopic pupil diameter <= 3.5 mm in each eye

Exclusion Criteria:

* Allergy to phenylephrine hydrochloride, tropicamide, or benzalkonium chloride
* History of benign prostatic hyperplasia
* Use of a benzodiazepine, monoamine oxidase inhibitor, tricyclic antidepressant, anticonvulsant, or cholinergic drug
* History of closed-angle glaucoma
* Anatomically narrow anterior chamber angles
* Ocular surgery or laser treatment of any kind
* History of chronic or acute uveitis
* History of traumatic iritis or hyphema
* History of traumatic mydriasis or angle recession
* History of heterochromia
* Irregularly-shaped pupil secondary to ocular trauma or congenital defect.
* History of neurogenic pupil disorder
* History of anterior chamber intraocular lens (IOL) or iris-fixated IOL
* History of iris surgery, iris atrophy, or iris-cornea apposition/touch
* Unwilling or unable to discontinue use of contact lenses at treatment visits.
* Current active eye disease for which topical or systemic ophthalmic medication is necessary, except for dry eye disease managed using artificial tears.
* Presence of a severe/serious ocular condition, or any other unstable medical condition that, in the Investigator's opinion, may preclude study treatment and/or follow-up
* Pregnancy or lactation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsontcho Ianchulev, MD, MPH, Study Director — Eyenovia Inc.
Locations (2):
- United States (2):
  - Keystone Research, Austin, Texas
  - R&R Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 76 patients signed the study informed consent form and were screened for eligibility between November 19, 2018 and December 14, 2018 at clinical research centers located in San Antonio and Austin, Texas.
Pre-assignment Details: 70 of the 76 participants enrolled initiated study treatment. Of those who did not initiate treatment, 4 failed to meet all study eligibility criteria and 2 were exited after screening (before treatment) because the required number of subjects had initiated treatment.
Units Other Than Participants: eyes
Groups:
- 1-TR/PE, 2-Placebo, 3-Placebo: Participants were administered the assigned treatment in each eye on separate days in the following order: 1st Treatment Day: Tropicamide 1%/Phenylephrine 2.5%, 2nd Treatment Day: Placebo, 3rd Treatment Day: Placebo. Each treatment was administered with the Optejet microdose dispenser.
- 1-Placebo, 2-Placebo, 3-TR/PE: Participants were administered the assigned treatment in each eye on separate days in the following order: 1st Treatment Day: Placebo, 2nd Treatment Day: Placebo, 3rd Treatment Day: Tropicamide 1%/Placebo 2.5%. Each treatment was administered with the Optejet microdose dispenser.
Period: Overall Study
Arm/Group | 1-TR/PE, 2-Placebo, 3-Placebo | 1-Placebo, 2-Placebo, 3-TR/PE
Started | 37; 74 eyes | 33; 66 eyes
Completed | 37; 74 eyes | 32; 64 eyes
Not Completed | 0; 0 eyes | 1; 2 eyes
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were administered the assigned treatments on 3 separate days (treatment administration sequence was randomized).
Arm/Group | All Participants
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (14.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 62
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 70
Iris Color Category [Count of Participants; unit: Participants] — Dark = Brown/black irides Light = All other colors
  Participants
    Dark | 50
    Light | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Pupil Diameter From Baseline
Description: Difference in 35-minute pupil diameter vs. baseline measured using pupillometry in highly photopic conditions.
  Pupil diameter is reported in millimeters. For the change in pupil diameter, larger measurements indicate a better outcome.
Time Frame: 35 minutes after initial dose
Population: Per-protocol population (participants who completed all planned assessments without a major protocol deviation)
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: eyes
Groups:
- TR/PE - Right Eye: Tropicamide 1%/Phenylephrine 2.5% ophthalmic solution administered to the right eye with the Optejet microdose dispenser
- TR/PE - Left Eye: Tropicamide 1%/Phenylephrine 2.5% ophthalmic solution administered to the left eye with the Optejet microdose dispenser.
- Placebo - Right Eye: Placebo ophthalmic solution administered to the right eye with the Optejet microdose dispenser
- Placebo - Left Eye: Placebo ophthalmic solution administered to the left eye with the Optejet microdose dispenser
Arm/Group | TR/PE - Right Eye | TR/PE - Left Eye | Placebo - Right Eye | Placebo - Left Eye
Number analyzed (Participants) | 69 | 69 | 69 | 69
Number analyzed (eyes) | 69 | 69 | 69 | 69
millimeters
  Change in 35-minute pupil diameter | 4.747 (0.7301) | 4.779 (0.8032) | 0.134 (0.4972) | 0.032 (0.4983)
  Baseline pupil diameter | 2.597 (0.4784) | 2.524 (0.4802) | 2.632 (0.5202) | 2.559 (0.4666)
  35-minutes pupil diameter | 7.344 (0.7981) | 7.304 (0.8264) | 2.766 (0.6598) | 2.590 (0.5892)

2. Other Pre Specified Outcome: Proportion of Eyes Achieving Pupil Diameter 6.0 mm or Larger After Receipt of Each Medication
Description: The percent of eyes with pupil diameter 6.0 mm or larger as measured using pupillometry in highly photopic conditions. As this is a cross-over study, each of the 69 participants received each medication. Data is reported separately for the right and left eyes of the 69 participants. A higher percentage indicates a better outcome.
Time Frame: 35 minutes after initial dose
Population: Per-protocol population (participants who completed all planned assessments without a major protocol deviation)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | TR/PE - Right Eye | TR/PE - Left Eye | Placebo - Right Eye | Placebo - Left Eye
Number analyzed (Participants) | 69 | 69 | 69 | 69
Number analyzed (eyes) | 69 | 69 | 69 | 69
percentage of eyes | 92.8 | 94.2 | 0 | 0

3. Other Pre Specified Outcome: Proportion of Eyes Achieving Pupil Diameter 7.0 mm or Larger After Receipt of Each Medication
Description: The percent of eyes with pupil diameter 7.0 mm or larger as measured using pupillometry in highly photopic conditions. As this is a cross-over study, each of the 69 participants received each solution. Data is reported separately for the right and left eyes of the 69 participants. A higher percentage indicates a better outcome.
Time Frame: 35 minutes after initial dose
Population: Per-protocol population (participants who completed all planned assessments without a major protocol deviation)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | TR/PE - Right Eye | TR/PE - Left Eye | Placebo - Right Eye | Placebo - Left Eye
Number analyzed (Participants) | 69 | 69 | 69 | 69
Number analyzed (eyes) | 69 | 69 | 69 | 69
percentage of eyes | 69.6 | 68.1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over each participant's study participation period, which was a maximum of 14 days.
Groups:
- Tropicamide/Phenylephrine: Tropicamide 1%/Phenylephrine 2.5% ophthalmic solution administered with the Optejet microdose dispenser
- Placebo: Placebo ophthalmic solution administered with the Optejet microdose dispenser
Arm/Group | Tropicamide/Phenylephrine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/70
Other Adverse Events (participants affected / at risk) | 2/69 | 0/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tropicamide/Phenylephrine (N=69) | Placebo (N=70)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Instillation site pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT03751098/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03751098/SAP_001.pdf
  • Informed Consent Form (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT03751098/ICF_002.pdf